CLINICAL TRIAL: NCT05368051
Title: Multi-omics Model Predicts Efficacy of Preoperative Neoadjuvant Chemoradiotherapy Combined PD-1 Antibody Therapy for Locally Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Other Study IDs: BFH-MMCRP
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- long course radiotherapy + capecitabine + PD-1 monoclonal antibody: long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations in patients with locally advanced rectal cancer
  Interventions: Combination Product: long course radiotherapy + capecitabine + PD-1 monoclonal antibody

INTERVENTIONS:
Combination Product: long course radiotherapy + capecitabine + PD-1 monoclonal antibody — long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations in patients with locally advanced rectal cancer

SUMMARY:
The purpose of this clinical research is to establish a multi-omics model based on genomics，transcriptomics，gut microbiota in predicting pathologic response after neoadjuvant chemoradiotherapy combined PD-1 antibody given to patients with locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been fully aware of the content of this study and signed the informed consent voluntarily;
* Patients with rectal cancers must satisfied all the following conditions: Stage II/III LARC (cT1-3N1-2M0)；Tumor distal location ≤ 7 cm from anal verge (MRI diagnosed);
* Patients regardless of gender with aged ≥18 years and ECOG score of 0 or 1;
* Physical and viscera function of patients can withstand major abdominal surgery;
* Patients are willing and able to follow the study protocol during the study;
* Patients give consent to the use of blood and pathological specimens for study;
* Within 28 days prior to enrolment, we must confirm a negative serological pregnancy test for child-bearing age women and they agree to use effective contraception for the duration of drug use and for 60 days after the last dose.

Exclusion Criteria:

* Patients have a present or previous active malignancy except the diagnosis of rectal cancer this time;
* Patients underwent major surgery within 4 weeks prior to study treatment;
* Patients have any condition affects the absorption of capecitabine through gastrointestinal tract;
* Patients have severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
* Patients who are allergic to any of the ingredients under study;
* Patients with severe concomitant diseases with estimated survival ≤ 5 years;
* Patients with present or previous moderate or severe liver and kidney damage presently or previously;
* Patients have received other study medications or any immunotherapy currently or in the past;
* Patients preparing for or previously received organ or bone marrow transplant;
* Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of study therapy;
* Patients with congenital or acquired immune deficiency (such as HIV infection);
* If patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the investigator will determine whether the clinical severity prevents the signing of informed consent or affects the patient's oral medication compliance;
* Patients with other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment and severe laboratory examination abnormalities.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mid to low LARC
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 1 year
  All the enrolled patients will receive total mesorectal excision (TME) 7-9 weeks after the end of long course radiotherapy. The rectal specimens will be evaluated by the pathologists who are experienced on the rectal cancer diagnosis according to the 1997 Dworak grading system. The rectal cancer will be classified into 5 grades. Grade 0-3 will be considered as non-pCR while grade 4 represent pCR.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Yao, Dr, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma J, Sun S, Cheng X, Meng C, Zhao H, Fu W, Gao Y, Ma L, Yang Z, Yao H, Su J. Unraveling the role of gut microbiome in predicting adverse events in neoadjuvant therapy for rectal cancer. Hum Vaccin Immunother. 2024 Dec 31;20(1):2430087. doi: 10.1080/21645515.2024.2430087. Epub 2024 Dec 2. PMID 39623529